CLINICAL TRIAL: NCT03985657
Title: Sleep Disordered Breathing in Marfan Syndrome: Susceptibility and Hemodynamics
Brief Title: Hemodynamics Response to Upper Airway Obstruction in Marfan Syndrome
Acronym: MSB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: The Marfan Foundation (Other); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IRB00157403
Record Dates: First submitted 2019-06-11; First posted 2019-06-14 (Actual); Results first posted 2020-12-28 (Actual); Last update posted 2020-12-28 (Actual); Status verified 2020-12

CONDITIONS: Sleep-disordered Breathing; Snoring
MeSH Terms: conditions — Sleep Apnea Syndromes; Snoring

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to a Baseline polysomnography and CPAP polysomnography in a randomized fashion. Participants will then be switched to the second polysomnography within 14 days of the first. The baseline polysomnography represents the exposure to sleep disordered breathing and the CPAP polysomnography represents the relief of the exposure. Markers of hemodynamic stress will be assessed in the morning after both studies.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Baseline Sleep Study (Active Comparator): Baseline sleep polysomnography will involve the collection of electroencephalogram, electromyogram, electrocardiogram, airflow, heart rate, blood pressure, and pleural pressure during sleep with no CPAP. Participants in this arm would switch to CPAP within one week of the study.
  Interventions: Device: CPAP
- CPAP Sleep Study (Experimental): Participants will be treated with continuous positive airway pressure to relieve sleep-disordered breathing. Participants in this arm would switch to Baseline study within one week of the study.
  Interventions: Device: CPAP

INTERVENTIONS:
Device: CPAP — Continuous positive airway pressure (CPAP). Room air at pressures between 6-8 centimeters of water (cmH2O) delivered via heated humidified tubing and a nasal mask.

SUMMARY:
Upper airway obstruction (UAO) is an unrecognized source of hemodynamic stress that may contribute to aortic adverse events in persons with Marfan Syndrome (MFS). UAO occurs during snoring and sleep apnea and is characterized by repetitive partial or complete obstruction of the upper airway during sleep. These obstructive breathing events lead to intermittent surges in blood pressure (BP) REF and large decreases in pleural pressure (Pes), thereby increasing the trans-mural aortic pressure (TMP) and imposing mechanical stress on the aorta during sleep. Although UAO is known to increase mechanical stress on the aorta, the magnitude of the increase is not known for persons with MFS.

In this project, therefore, the investigators will also examine the changes in Pes and BP responses in periods of obstructed breathing and compare the diurnal markers or vascular stress between Baseline and CPAP studies in MFS persons.

DETAILED DESCRIPTION:
Research Objective/Significance:

Specific Aim 1a: To quantify the Pes and BP during periods with and without UAO during sleep in persons with MFS.

Specific Aim 1b: To examine the effect of CPAP treatment of UAO on Pes and BP in MFS persons.

Specific Aim 2: To examine the effect of CPAP treatment of UAO on daytime markers of hemodynamic stress (augmentation index, reactive hyperemia index) in MFS persons.

Primary Outcomes:

* Overnight measure of hemodynamic stress (blood pressure, pleural pressure swings)

Secondary Outcomes:

* Changes in diurnal markers of hemodynamic stress (augmentation index, reactive hyperemia index)

ELIGIBILITY:
Inclusion Criteria:

People with Marfan syndrome.

* Age ≥ 18yrs
* Able and willing to provide informed consent
* Willing to sleep connected to research apparatus

Exclusion Criteria:

* Unstable cardiovascular disease (CHF, myocardial infarction or revascularization procedures, and unstable arrhythmias)
* Uncontrolled hypertension (BP > 190/110)
* Underlying obstructive or other intrinsic lung disease
* Renal failure on dialysis
* Cirrhosis
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2018-06-06 (Actual); Primary Completion 2019-12-06 (Actual); Study Completion 2019-12-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mudiaga Sowho, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 193 persons with Marfan syndrome were screened. Persons were recruited from the Johns Hopkins Marfan Clinic and the external Marfan Community via the Marfan foundation. Inclusion was based on a clinical diagnosis of Marfan syndrome (Ghent Criteria) or genetic testing. Persons were excluded if they had any chronic lung disease, other sleep disorders aside from sleep apnea, were on blood thinners, or had uncontrolled blood pressure. Recruitment occurred between 09/2018 and 11/2019.
Groups:
- Baseline Sleep Study: Baseline sleep polysomnography involved the monitoring of electroencephalogram, electromyogram, electrocardiogram, airflow, heart rate, blood pressure, and pleural pressure during sleep with no CPAP. Participants in this arm would switch to CPAP within one week of the Baseline Sleep Study.
- CPAP Sleep Study: In a randomized cross-over fashion, participants were treated with continuous positive airway pressure (CPAP) on a separate night. Room air at pressures between 6-9 centimeters of water (cmH2O) were delivered via heated humidified tubing and a nasal mask. Participants in this arm would switch to Baseline Sleep Study within one week of the CPAP Sleep Study.
Period: Intervention 1 (One Night)
Arm/Group | Baseline Sleep Study | CPAP Sleep Study
Started | 20 | 11
Completed | 20 | 10
Not Completed | 0 | 1
Period: Washout (Up to 1 Week)
Arm/Group | Baseline Sleep Study | CPAP Sleep Study
Started | 20 | 10
Completed | 20 | 10
Not Completed | 0 | 0
Period: Intervention 2 (One Night)
Arm/Group | Baseline Sleep Study | CPAP Sleep Study
Started | 20 | 10
Completed | 20 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: All participants enrolled in this study.
Arm/Group | All Participants
Number analyzed (Participants) | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.5 (15.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 14
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 31

OUTCOME MEASURES:

1. Primary Outcome: Pleural Pressure (Pes)
Description: Pleural pressure (Pes) in mmHg monitored using an esophageal catheter.
Time Frame: Overnight on both CPAP and No CPAP nights
Population: Participants with upper airway obstruction (apneas, hypopneas, and flow limitation) during the Baseline sleep study, who had pleural pressure and blood pressure data collected during both Baseline and CPAP sleep studies.
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Baseline Sleep Study: Baseline sleep polysomnography will involve the collection of electroencephalogram, electromyogram, electrocardiogram, airflow, heart rate, blood pressure, and pleural pressure during sleep with no CPAP.
- CPAP Sleep Study: Participants will be treated with continuous positive airway pressure to relieve sleep-disordered breathing. CPAP: Continuous positive airway pressure (CPAP). Room air at pressures between 6-8 centimeters of water (cmH2O) delivered via heated humidified tubing and a nasal mask.
Arm/Group | Baseline Sleep Study | CPAP Sleep Study
Number analyzed (Participants) | 10 | 10
mmHg | 9.3 (3.4) | 4.4 (1.6)

2. Primary Outcome: Mean Arterial Blood Pressure (MAP)
Description: Continuous blood pressure monitored using a non-invasive finger cuff. Data captured in mmHg.
Time Frame: Overnight on both Baseline and CPAP studies
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Baseline Sleep Study | CPAP Sleep Study
Number analyzed (Participants) | 10 | 10
mmHg | 93.8 (14.0) | 88.3 (12.4)

3. Secondary Outcome: Augmentation Index (AI)
Description: The AI (measured as "percentage of pulse pressure") was assessed in the morning after both Baseline and CPAP studies. It is a measure of arterial stiffness that represents the degree of and can range from -10% to +10% in healthy individuals, with values generally higher in females and increases with age.
Time Frame: 15 minutes in the morning post Baseline and CPAP studies
Population: Participants with adequate sleep time (>2hrs) on both Baseline and CPAP studies and AI measurements after both Baseline and CPAP studies.
Measure: Mean (Standard Error); unit: percentage of pulse pressure
Arm/Group | Baseline Sleep Study | CPAP Sleep Study
Number analyzed (Participants) | 28 | 28
percentage of pulse pressure | 11.0 (3.8) | 2.4 (3.7)

4. Secondary Outcome: Reactive Hyperemia Index (RHI)
Description: The RHI is a measure of endothelial function that was measured in the morning after both Baseline and CPAP studies. It is unitless and scored on a range of 1 to 3 in healthy individuals with lower values indicating poor endothelial function.
Time Frame: 15 minutes
Population: Participants with adequate sleep time (>2hrs) on both Baseline and CPAP studies and morning RHI measurements after both Baseline and CPAP studies.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Baseline Sleep Study | CPAP Sleep Study
Number analyzed (Participants) | 26 | 26
score on a scale | 2.2 (0.1) | 2.2 (0.2)

ADVERSE EVENTS:
Time Frame: Over the two night sessions.
Groups:
- Baseline Sleep Study: Baseline sleep polysomnography involved the monitoring of electroencephalogram, electromyogram, electrocardiogram, airflow, heart rate, blood pressure, and pleural pressure during sleep with no CPAP.
- CPAP Sleep Study: Participants were treated with continuous positive airway pressure (CPAP) on a separate night. Room air at pressures between 6-9 centimeters of water (cmH2O) were delivered via heated humidified tubing and a nasal mask.
Arm/Group | Baseline Sleep Study | CPAP Sleep Study
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/31
Other Adverse Events (participants affected / at risk) | 0/30 | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-16): https://cdn.clinicaltrials.gov/large-docs/57/NCT03985657/Prot_SAP_000.pdf